CLINICAL TRIAL: NCT00651040
Title: A Prospective, Randomised, Assessor-blind, Multicenter Study of Efficacy and Safety of Combined Treatment of Methotrexate + Glucocorticoids Versus Glucocorticoids Alone in Patients With Polymyositis and Dermatomyositis.
Brief Title: Combined Treatment of Methotrexate + Glucocorticoids Versus Glucocorticoids Alone in Patients With PM and DM
Acronym: Prometheus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Rheumatology, Prague (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3401
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Polymyositis; Dermatomyositis
Keywords: Polymyositis; Dermatomyositis; Glucocorticoids; Methotrexate
MeSH Terms: conditions — Polymyositis; Dermatomyositis | interventions — Prednisone; Prednisolone; Methotrexate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednison (Active Comparator): Prednisone will be administered orally, initially at 1.0 mg/kg/day dosage and then tapered gradually equally in the two arms.
  ARM 1 has only Prednisone
  Interventions: Drug: Prednisone
- Prednison + methotrexate (Active Comparator): MTX will be administered orally (in case of oral intolerance intramusculary (i.m.)), once weekly for 48 weeks. There will be a clinically oriented dose escalation starting from 10 up to 20-25 mg of MTX. Five to ten mg of folic acid will be given 24 hours after each methotrexate dose.
  Interventions: Drug: Prednisone; Drug: Methotrexate

INTERVENTIONS:
Drug: Prednisone — Prednisone will be administered orally, initially at 1.0 mg/kg/day dosage and then tapered gradually equally in the two arms
  Other Names: Prednisolone
Drug: Methotrexate — MTX will be administered orally (in case of oral intolerance intramusculary (i.m.)), once weekly for 48 weeks. There will be a clinically oriented dose escalation starting from 10 up to 20-25 mg of MTX. Five to ten mg of folic acid will be given 24 hours after each methotrexate dose.
  Arms: Prednison + methotrexate

SUMMARY:
Therapeutical trial in patients with idiopathic polymyositis (PM) and dermatomyositis (DM) is proposed. The study will investigate the safety and efficacy of combined methotrexate (MTX) + glucocorticoids (GC) treatment compared with GC alone.

This will be a randomised, open-label, assessor-blind, international multicenter trial, performed in several European centres interested in research on inflammatory myopathies (IIM).

A total number of 50 patients with PM/DM will be randomised into two groups (1: MTX+ GC and 2: GC only). Patients will be equally distributed between the two groups providing 25 patients per treatment arm. The randomisation will be based on random numbers generated by a computer program. After being enrolled in the study, the patients will receive 12 months of therapy followed by a 12-month follow-up period.

The primary endpoint is the total dose of GC ( in mg/kg weight), which will be administered for 12 months between baseline and the end of treatment.

There are several of secondary objectives, which will be pursued during and after the trial. Disease activity and damage will be prospectively assessed by tools for myositis disease activity (MYOACT and MITAX) and for myositis damage (MYODAM and MDI), global assessment of activity and damage by patients and by physician, muscle endurance, muscle strength by manual muscle testing, enzyme levels, GC related side effects, functional ability measured by HAQ, quality of life by SF-36, and number of patients with treatment failures. The other aims will also include (i) search for reliable prognostic parameters in the further prognosis of patients with PM/DM and (ii) studies on the pathogenic aspects of IIM. The investigations of serum, lymphocytes, muscle tissue and MRI will be organized. DNA and RNA will be stored for future genetic studies.

Patients with definite or probable PM or DM diagnosed according to diagnostic criteria will be enrolled. They will have disease activity that according to physician's own judgement requires high dose immunosuppressive treatment (based on clinical assessment of weakness, elevation of muscle enzymes and, if available, on magnetic resonance imaging findings). Patients should be previously untreated with the exception of GC treatment up to 8 weeks.

Patients with other than primary idiopathic PM or DM, such as drug-induced myositis, myositis in association with other connective tissue disease, inclusion body myositis, malignancy related myositis, and juvenile DM will be excluded.

All patients will start with prednisone 1 mg/kg/day and the dose will be tapered if patients meet definition of improvement, which has been proposed by IMACS group. MTX will be administered orally, once weekly, with a starting dose 10 mg. This will be increased gradually to 25 mg/week if tolerated by week 5. Patients will be first assessed after 2 weeks and than monthly for a period of 48 weeks. There will be a follow-up after a further 1 year in order to find out the impact of the early treatment on the long-term disease outcome.

All efficacy analyses will be performed using intention-to-treat population (ITT). In addition, the primary and secondary variables will be analysed using the per-protocol population, which will contain all patients in the ITT population, who also reached Week 48 without any major protocol violations. The safety population, which will contain any patient who received at least one dose of study drug, will be used for all safety analyses.

DETAILED DESCRIPTION:
Clinical trial:

A prospective, randomized, assessor- blind, multicenter study of safety and efficacy of combined treatment of methotrexate and glucocorticoids versus glucocorticoids alone in patients with polymyositis and dermatomyositis

Tested investigational medicinal product: Methotrexate (Methotrexatum dinatricum 2,5 mg tbl.).

Mechanism of Action: Methotrexate inhibits dihydrofolic acid reductase. Dihydrofolates must be reduced to tetrahydrofolates by this enzyme before they can be utilized as carriers of one-carbon groups in the synthesis of purine nucleotides and thymidylate. Therefore, methotrexate interferes with DNA synthesis, repair, and cellular replication. Actively proliferating tissues such as malignant cells, bone marrow, fetal cells, buccal and intestinal mucosa, and cells of the urinary bladder are in general more sensitive to this effect of methotrexate.

Comparator : Prednison (Prednisonum 20 mg tbl.)

Mechanism of Action: Glucocorticoids are naturally occurring hormones that prevent or suppress inflammation and immune responses when administered at pharmacological doses. At a molecular level, unbound glucocorticoids readily cross cell membranes and bind with high affinity to specific cytoplasmic receptors. This binding induces a response by modifying transcription and, ultimately protein synthesis to achieve the steroid's intended action. Such actions may include: inhibition of leukocyte infiltration at the site of inflammation, interference in the function of mediators of inflammatory response, and suppression of humoral immune responses. Some of the net effects include reduction in edema or scar tissue, as well as a general suppression in immune response. The degree of clinical effect is normally related to the dose administered. The antiinflammatory actions of corticosteroids are thought to involve phospholipase A2 inhibitory proteins, collectively called lipocortins. Lipocortins, in turn, control the biosynthesis of potent mediators of inflammation such as prostaglandins and leukotrienes by inhibiting the release of the precursor molecule arachidonic acid. Likewise, the numerous adverse effects related to corticosteroid use are usually related to the dose administered and the duration of therapy.

Number of patients in the trial:

* Total 50
* In this centre: 10

Summary:

The aim of the study is to determine the safety and efficacy of adding methotrexate (MTX) to glucocorticoids (GC) compared with glucocorticoid treatment alone in patients with inflammatory myopathies.

1. PM and DM are usually treated with glucocorticoids and immunosuppressive drugs. However, such treatment has not yet been studied thoroughly and properly evaluated in a randomized controlled trial. There are only few controlled studies of PM/DM management and all of them have been performed in small groups of patients. This will be the first randomized controlled trial with MTX
2. This clinical trial will assess efficacy MTX in patients with early PM/DM
3. Also long- term effect of treatment (MTX and glucocorticoids versus glucocorticoids) will be evaluated.
4. Inclusion criteria allow to follow up the consistent group of PM/DM patients.
5. In this trial the of newly developed tools for myositis disease activity will be used
6. The secondary objectives is to study pathogenic aspects of inflammatory myopathies.
7. The serum, DNA and RNA will be stored for future genetic studies and to study autoantibodies to search for prognostic markers.

Objectives:

The primary objective of the study is to determine the safety and efficacy of adding methotrexate (MTX) to glucocorticoids (GC) compared with glucocorticoid treatment alone in patients with inflammatory myopathies. The primary endpoint that will be measured is the total dose of glucocorticoids (in mg/kg weight) administered between baseline and the end of treatment.

The secondary objectives are:

1. Assessment of disease activity and damage [with the use of newly developed tools for myositis disease activity (MYOACT and MITAX) and myositis damage (MYODAM and MDI), as well as by global assessment of activity and damage by patients and by physician.
2. Muscle strength by manual muscle testing
3. Muscle endurance
4. Muscle enzyme levels
5. Glucocorticoid related side-effects
6. Final glucocorticoid dose
7. Disability index by HAQ
8. Quality of life by SF-36
9. Number of patients with treatment failures
10. Search for reliable prognostic parameters in the further prognosis of patients with inflammatory myopathies.

Study of the pathogenic aspects of inflammatory myopathies. Therefore investigations of serum, lymphocytes, muscle tissue and MRI will be organized. DNA and RNA will be stored for future genetic studies.

Study design.

This will be a randomized, assessor-blinded, multicenter, international study. After being enrolled in the study, the patients will receive 48 weeks of therapy followed by a 12-month follow-up period.

A total number of 50 patients with polymyositis/dermatomyositis are planned to be randomized. These will be equally distributed between the two groups providing 25 patients per treatment arm. Patients will be randomized on the basis of random numbers generated by a computer program.

Indication:

Treatment of active polymyositis and dermatomyositis

Evaluations.

Efficacy. The efficacy will be assessed by fulfillment of definition of improvement at every visit and treatment taper with glucocorticoids. Overall efficacy will be assessed by measurement of disease activity (MITAX, MYOACT), disease damage (MDI, MYODAM), global patient's and physician's assessments, manual muscle strength test, functional muscle test2, health assessment questionnaire (HAQ), and SF36.

Safety.

The safety will be assessed at every visit by clinical and laboratory examinations. Specifically, clinical assessment will include physical examination, vital signs, muscle function index, manual muscle strength test, MYOACT, MITAX, MYODAM, MDI, HAQ and global assessment of activity and damage by physician and patient.

Laboratory assessments will include complete blood count, blood chemistry including SGOT (AST), SGPT (ALT), Na, K, creatinine, LDH, CK, CRP and urine pregnancy test if required by local practice.

In patients with pulmonary alveolitis or interstitial fibrosis at the start of the study - HRCT should be performed. If significant progress of pulmonary infiltrate will occur, this is considered to be treatment failure and patient will be treated according to standard approach.

Pulmonary toxicity from methotrexate can be suspected in patients with sudden onset of nonproductive cough with dyspnea. HRCT should be performed. If there are no other obvious reasons for these symptoms methotrexate should be discontinued.

If nausea after methotrexate occurs, try to divide the dose or give antinauseous drug. If there are still unacceptable gastrointestinal side effects, parenteral methotrexate administration can be considered.

Patient selection

Inclusion criteria:

1. Age between 18 - 80 years.
2. Patients with definite or probable polymyositis or dermatomyositis diagnosed according to diagnostic criteria (9, 10) (Appendix 1)
3. Physician's own judgment of the disease activity that requires high dose immunosuppressive treatment (based on clinical assessment of weakness, elevation of muscle enzymes and, if available, on magnetic resonance imaging findings).
4. Previously untreated patients with the exception of glucocorticoid treatment up to 8 weeks
5. Signed informed consent.

Exclusion criteria:

1. Treatment with any immunosuppressive drug prior the study start.
2. Treatment with glucocorticoids (> 20 mg of Prednisone or equivalent) more than 8 weeks prior to study start.
3. Drug induced myositis.
4. Polymyositis and dermatomyositis in association with other connective tissue disease.
5. Inclusion body myositis.
6. Patients with immunodeficiency syndrome.
7. Pregnancy and lactation.
8. Fertile women not using adequate contraception during the study, women planning to have children during the study course or 12 months after the end of the study.
9. Malignancy.
10. Juvenile dermatomyositis.
11. Uncontrolled, clinically significant hematological, cardiovascular, pulmonary, endocrine, metabolic, gastrointestinal, hepatic or renal disease, which according to physician's consideration would interfere with high dose glucocorticoid and immunosuppressive treatment or would prevent to follow the treatment protocol.
12. Severe infection.
13. History of drug or alcohol abuse within the previous 6 months.
14. Patients known to be HIV positive.
15. Known hypersensitivity to methotrexate.

Withdrawal from study.

Patients will be withdrawn from the study due to following reasons:

1. non-compliance with the study protocol
2. positive pregnancy for female patients test during the course of the study
3. if worsening occurs
4. use of prohibited concomitant treatment
5. any adverse event which in the investigator´s opinion may compromise health of a study subject

Treatment MTX will be administered orally (in case of oral intolerance intramusculary (i.m.)), once weekly for 48 weeks. There will be a clinically oriented dose escalation starting from 10 up to 20-25 mg of MTX. Five to ten mg of folic acid will be given 24 hours after each methotrexate dose.

Prednisone will be administered orally, initially at 1.0 mg/kg/day dosage and then tapered gradually equally in the two arms

Concomitant medication and treatment:

Recommended medication- Five to ten mg of folic acid will be given 24 hours after each methotrexate dose.

Prohibited medication: Other immunosuppressive agents are not allowed. All other medication is allowed at the discretion of the investigator.

Study flowchart Controls and visits will be organized: Day 0 (Baseline), in the 2.week, in the 1.,2., 3. 4., 5., 6., 7., 8., 9. 10. 11. and 12.month (Termination visit), than one year Follow-up

Statistics.

Summary statistics of the baseline characteristics will be tabulated by treatment group.

The main population for evaluation will be the ITT (intent- to-treat) population. Summary statistics (N, mean, standard deviation, median, minimum and maximum) will be presented for each treatment group by visit for the continuous variables. For the categorical variables N and % will be presented for each treatment group at endpoint.

A total number of 50 patients with polymyositis/dermatomyositis are planned to be randomized. These will be equally distributed between the two groups providing 25 patients per treatment arm. Two-sided tests at the 5% level of significance The primary endpoint that will be measured is the total dose of glucocorticoids (in mg/kg weight) administered between baseline and end of treatment.

Between treatment differences will be tested using parametric (t-test) and non-parametric tests (Mann-Whitney test).

The secondary efficacy variables are disease activity and damage measures, which will be assessed by myositis disease activity assessment tools (MYOACT and MITAX), myositis damage tools (MYODAM, MDI), and global assessment of activity and damage by patients and by physician The continuous secondary variables at endpoint will be tested for treatment differences using parametric (t-test, ANOVA) and non-parametric tests (Mann-Whitney test, Kruskal-Wallis ANOVA).

In the event that at the time of statistical analysis any of the model assumptions are not met data transformations or alternative methods of analysis will be performed as appropriate.

The categorical secondary efficacy variables will be tested for treatment differences using Fischer's exact test.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 - 80 years.
2. Patients with definite or probable polymyositis or dermatomyositis diagnosed according to diagnostic criteria (9, 10) (Appendix 1)
3. Physician's own judgment of the disease activity that requires high dose immunosuppressive treatment (based on clinical assessment of weakness, elevation of muscle enzymes and, if available, on magnetic resonance imaging findings).
4. Previously untreated patients with the exception of glucocorticoid treatment up to 8 weeks
5. Signed informed consent.

Exclusion Criteria:

1. Treatment with any immunosuppressive drug prior the study start.
2. Treatment with glucocorticoids (> 20 mg of Prednisone or equivalent) more than 8 weeks prior to study start.
3. Drug induced myositis.
4. Polymyositis and dermatomyositis in association with other connective tissue disease.
5. Inclusion body myositis.
6. Patients with immunodeficiency syndrome.
7. Pregnancy and lactation.
8. Fertile women not using adequate contraception during the study, women planning to have children during the study course or 12 months after the end of the study.
9. Malignancy.
10. Juvenile dermatomyositis.
11. Uncontrolled, clinically significant hematological, cardiovascular, pulmonary, endocrine, metabolic, gastrointestinal, hepatic or renal disease, which according to physician's consideration would interfere with high dose glucocorticoid and immunosuppressive treatment or would prevent to follow the treatment protocol.
12. Severe infection.
13. History of drug or alcohol abuse within the previous 6 months.
14. Patients known to be HIV positive.
15. Known hypersensitivity to methotrexate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Vencovsky, prof. MD., Principal Investigator — Institute of Rheumatology, Prague
Locations (1):
- Revmatologicky ustav, Prague, Czechia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial has reached 62% of planned recruitment (31 patients randomized).
Groups:
- 1Prednison: Prednisone will be administered orally, initially at 1.0 mg/kg/day dosage and then tapered gradually equally in the two arms.
  ARM 1 has only Prednisone
  Prednisone: Prednisone will be administered orally, initially at 1.0 mg/kg/day dosage and then tapered gradually equally in the two arms
- 2Prednison MTX: MTX will be administered orally (in case of oral intolerance intramusculary (i.m.)), once weekly for 48 weeks. There will be a clinically oriented dose escalation starting from 10 up to 20-25 mg of MTX. Five to ten mg of folic acid will be given 24 hours after each methotrexate dose.
  Methotrexate: MTX will be administered orally (in case of oral intolerance intramusculary (i.m.)), once weekly for 48 weeks. There will be a clinically oriented dose escalation starting from 10 up to 20-25 mg of MTX. Five to ten mg of folic acid will be given 24 hours after each methotrexate dose.
Period: Overall Study
Arm/Group | 1Prednison | 2Prednison MTX
Started | 16 | 15
Completed | 13 | 14
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1Prednison | 2Prednison MTX | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (14.4) | 53.5 (17.4) | 52.6 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  Czech Republic | 13 | 8 | 21
  Sweden | 3 | 1 | 4
  Switzerland | 0 | 4 | 4
  Hungary | 0 | 1 | 1
  Poland | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Total Dose of Glucocorticoids Administered Between Baseline and the End of Treatment.
Description: The primary endpoint which has benn measured was the total dose of glucocorticoids administered between baseline and the end of treatment.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mg/kg
Groups:
- Prednison1: Prednisone will be administered orally, initially at 1.0 mg/kg/day dosage and then tapered gradually equally in the two arms.
  ARM 1 has only Prednisone
  Prednisone: Prednisone will be administered orally, initially at 1.0 mg/kg/day dosage and then tapered gradually equally in the two arms
- Prednison Methotrexate 2: MTX will be administered orally (in case of oral intolerance intramusculary (i.m.)), once weekly for 48 weeks. There will be a clinically oriented dose escalation starting from 10 up to 20-25 mg of MTX. Five to ten mg of folic acid will be given 24 hours after each methotrexate dose.
  Methotrexate: MTX will be administered orally (in case of oral intolerance intramusculary (i.m.)), once weekly for 48 weeks. There will be a clinically oriented dose escalation starting from 10 up to 20-25 mg of MTX. Five to ten mg of folic acid will be given 24 hours after each methotrexate dose.
Arm/Group | Prednison1 | Prednison Methotrexate 2
Number analyzed (Participants) | 16 | 15
mg/kg | 124 (65.7) | 135 (45.2)

2. Secondary Outcome: Assessment of Disease Activity and Damage,Muscle Strength and Endurance, Enzyme Levels, Glucocorticoid Side-effects, Dose, HAQ,SF-36, Treatment Failures
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2016-12

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- 1 Prednison: Prednisone will be administered orally, initially at 1.0 mg/kg/day dosage and then tapered gradually equally in the two arms.
  ARM 1 has only Prednisone
  Prednisone: Prednisone will be administered orally, initially at 1.0 mg/kg/day dosage and then tapered gradually equally in the two arms
- 2 Prednison Methotrexate: MTX will be administered orally (in case of oral intolerance intramusculary (i.m.)), once weekly for 48 weeks. There will be a clinically oriented dose escalation starting from 10 up to 20-25 mg of MTX. Five to ten mg of folic acid will be given 24 hours after each methotrexate dose.
  Methotrexate: MTX will be administered orally (in case of oral intolerance intramusculary (i.m.)), once weekly for 48 weeks. There will be a clinically oriented dose escalation starting from 10 up to 20-25 mg of MTX. Five to ten mg of folic acid will be given 24 hours after each methotrexate dose.
Arm/Group | 1 Prednison | 2 Prednison Methotrexate
Serious Adverse Events (participants affected / at risk) | 4/16 | 5/15
Other Adverse Events (participants affected / at risk) | 14/16 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Prednison (N=16) | 2 Prednison Methotrexate (N=15)
tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
worsening of muscles (Musculoskeletal and connective tissue disorders) | 2 | 0
worsening of skin (Skin and subcutaneous tissue disorders) | 0 | 1
synkopa (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Prednison (N=16) | 2 Prednison Methotrexate (N=15)
infection (Infections and infestations) | 8 | 6
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 | 3
cardiovascular (Cardiac disorders) | 2 | 2
gastrointestinal (Gastrointestinal disorders) | 2 | 3
general (General disorders) | 3 | 3
endocrine (Endocrine disorders) | 2 | 0
neurological (Nervous system disorders) | 3 | 0
psychiatric (Psychiatric disorders) | 1 | 0
gynecological (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes